CLINICAL TRIAL: NCT03892135
Title: Representation and Medication Use in Juvenile Idiopathic Arthritis - RUMAJI
Brief Title: Representation and Medication Use in Juvenile Idiopathic Arthritis
Acronym: RUMAJI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Research department, unknowns, Strategic & innovation consulting, Paris (anthropologists) (Unknown); NORDIC pharma (funding) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0171
Record Dates: First submitted 2019-03-18; First posted 2019-03-27 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-03

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Role of parents, children and physician; Qualitative; Interview; Juvenile idiopathic arthritis; Adherence; mechanisms of adherence in juvenile idiopathic arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Interviews as Topic; Physicians

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Physicians: 3 paediatricians and 3 rheumatologists
  Interventions: Other: Interviews with Physicians
- Parents: Parents
  Interventions: Other: Interviews with parents of children with juvenile idiopathic arthritis
- Children: Children
  Interventions: Other: Interviews with children with juvenile idiopathic arthritis

INTERVENTIONS:
Other: Interviews with parents of children with juvenile idiopathic arthritis — Interviews with parents of children with juvenile idiopathic arthritis
  Groups: Parents
Other: Interviews with children with juvenile idiopathic arthritis — Interviews with children with juvenile idiopathic arthritis
  Groups: Children
Other: Interviews with Physicians — Interviews with Physicians
  Groups: Physicians

SUMMARY:
According to the International League of Associations for Rheumatology classification, Juvenile Idiopathic Arthritis (JIA) comprises a heterogeneous group of arthritis of unknown cause and with onset before 16 years of age, characterized by joint inflammation lasting for 6 or more weeks. Few studies exist regarding the care experience of children affected by this rheumatic condition. On the other hand, methotrexate and biologics constitute the primary treatment for children with JIA. As with adults undergoing the same treatment, adherence is critical. Difficulties for children to take the drugs have been reported. Notwithstanding, if adherence promotion in pediatric chronic conditions has been the subject of recommendations with regard to care management, the investigators lack information to understand the grounds for adherence specifically in JIA. In order to understand and decipher the parent-child adherence mechanisms and practices, the RUMAJI study will be conducted. Indeed, improving the relational approach between children and their caregivers as well as unrestricted drug adherence involves researching and understanding how appropriation of the disease and treatment could be achieved.

ELIGIBILITY:
Inclusion criteria:

* all JIA forms
* all treatment type (NSAIDs, MTX, bDMARDs)

Exclusion criteria:

- none

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with JIA and their parents
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Interview with parents | 1 day
  Interview with parents to learn about role of parents in the management of juvenile idiopathic arthritis in their children

SECONDARY OUTCOMES:
Interview with children | 1 day
  Interview with children to learn about role of children in the management of their juvenile idiopathic arthritis
Interview with physicians | 1 day
  Interview with physicians to learn about role of physicians in the management of juvenile idiopathic arthritis

CONTACTS AND LOCATIONS:
Overall Officials: Jean-David COHEN, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC